CLINICAL TRIAL: NCT04738201
Title: Investigation of Clinical Effects of a Proprioceptive Thumb Exercises Program in Patients With Carpometacarpal Joint Osteoarthritis: A Randomized Clinical Trial
Brief Title: Proprioceptive Thumb Exercises Program in Patients With Carpometacarpal Joint Osteoarthritis
Acronym: thumb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Raquel Cantero-Téllez, Principal Investigator, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020
Record Dates: First submitted 2020-11-02; First posted 2021-02-04 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Thumb Osteoarthritis
Keywords: Thumb pain; Thumb proprioception; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Thumb orthosis at night. Daily exercises program during 4 weeks grouped in 3 sets of 10 repetitions in absence of pain. Exercises will consisted of active - resistive exercises for the first dorsal interosseous (FDI) muscle, manual distraction of the CMC joint and relaxation of the adductor thumb muscle.
  Interventions: Other: Proprioceptive thumb exercises.
- Experimental group (Experimental): The experimental group will also carried out a proprioceptive exercise program divided in three phases of 2 weeks per phase.
  Interventions: Other: Proprioceptive thumb exercises.

INTERVENTIONS:
Other: Proprioceptive thumb exercises. — Exercises for recognition of thumb position and thumb force sense.

SUMMARY:
Osteoarthritis (OA) is a chronic and prevalent joint disorder with great impact on quality of life and high economic burden. Although a number of conservative therapies have proven to be effective for the management of hand OA, only modest treatment effects were reported for most individual interventions. The aim of the proposed study is to assess the effect of proprioceptive training on pain, function and sense perception in patients with carpometacarpal osteoarthritis (CMC OA).

DETAILED DESCRIPTION:
A randomized, controlled, single-center, double-blind, clinical trial, with 1:1 allocation ratio, will be carried out involving patients diagnosis of CMC joint OA grade 1-2 (aged 18 years and above). Both assessor and statistician will remained blinded. The research diagnostic criteria for carpometacarpal joint osteoarthritis will be used to assess all individuals who agree to participate. Based on the clinical and radiological findings, the participants will be classified by a rheumatology. Those with CMC OA grade 2-3 will be included in the study.

Standard conservative thumb CMC joint OA treatments will received for both the control and experimental groups for a period of 12 weeks. The experimental group will received a proprioceptive training program during the same intervention period, which will be conducted twice weekly (24 sessions).

The severity of pain with activity will be measured according to the visual analog scale (VAS). QuickDASH questionnaire will be used to measure upper extremity function. Patient's occupational performance will be measured with the Canadian Occupational Performance Measure (COPM) and proprioception with Joint position sense (JPS) testing. All outcome measures will be collected at baseline, immediately following the intervention at 4 weeks and at 12 weeks following the end of the intervention.

Participation in the study will be voluntary and patients will be included if they satisfied specific inclusion criteria.

All procedures will be follow in accordance with the ethical standards of the responsible committee on human experimentation (institutional and national) and with the Helsinki Declaration. All participants will sign a written informed consent in accordance with guidelines approved by the local ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of grade I, II or III thumb CMC joint OA in their dominant hand according to the Eaton Classification Stage
* Pain rating of 4/10 on the Visual Analogue Scale (VAS) during activities of daily living (ADLs) at the time of the therapy initial evaluation.
* The ability to read and understand the patient information sheets and exercises

Exclusion Criteria:

* Neurological disorder affecting the upper limb.
* Had received specific treatment for hand or thumb pain in the same limb in the last 6 months including an intra-articular joint injection to wrist, fingers, or thumb; - Fractures or a significant hand injury or previous surgery to the wrist or hand;
* Tenosynovitis and/or Dupuytren disease

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women over 60 diagnosis with CMC joint OA
Enrollment: 45 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Joint position Sense (JPS) | baseline-4 and 12 weeks
  Proprioception using active joint position sense (JPS) has been utilized in studies to establish a correlation between therapy intervention and proprioception. The target position of 30º CMC abduction will be selected. Joint angle will be measured using a standard clear plastic goniometer.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | baseline-4 and 12 weeks
  VAS has been shown to be a reliable and valid instrument for pain assessment which is used frequently for clinical and research purposes. It consists of a 10-cm line anchored at each end. The left-hand anchor reads 'no pain' and the right-hand anchor reads 'worst possible pain'; the patients marked a line to represent their pain level.
Quick dash | baseline-4 and 12 weeks
  The QuickDASH questionnaire will be used to measure upper extremity function. This tool consists of 11 items providing a total score ranging from 0 to 100 where 0 indicates no limitation and 100 suggests full disability. Eight items include questions about the ability of the patient to perform certain daily activities.
Canadian Occupational Performance Measure | baseline-4 and 12 weeks
  Patient's occupational performance will be measured with the Canadian Occupational Performance Measure (COPM). The COPM enables subjects to identify goals for hand therapy and engage in a subject-specific therapeutic process. It has been established that the COPM has good convergent validity and responsiveness for evaluating the relationship between patient self-perception and satisfaction for patients with CMC thumb OA .

CONTACTS AND LOCATIONS:
Locations (1):
- Raquel Cantero-Téllez, Málaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cantero-Tellez R, Perez-Cruzado D, Villafane JH, Garcia-Orza S, Naughton N, Valdes K. The Effect of Proprioception Training on Pain Intensity in Thumb Basal Joint Osteoarthritis: A Randomized Controlled Trial. Int J Environ Res Public Health. 2022 Mar 17;19(6):3592. doi: 10.3390/ijerph19063592. PMID 35329279